CLINICAL TRIAL: NCT06250127
Title: The Effectiveness of Modified 3D Printed Customized Facemask Appliance for Treatment of Class III Malocclusion: A Randomized Clinical Trial
Brief Title: The Effectiveness of Modified 3D Printed Customized Facemask Appliance for Treatment of Class III Malocclusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 882423
Record Dates: First submitted 2024-01-21; First posted 2024-02-08 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Jaw Protrusions
Keywords: Orthopedic appliance; Maxillary protraction; Petit facemask; Cl III malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding to treatment allocation is possible only for the outcomes assessor because the clinicians know the intervention. The trial documents will be labeled with ID number, which be used for participant identification and data collection without unmasking the allocation group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Conventional facemask) (Active Comparator): Conventional facemask appliance will be used for growing patients who have Cl. III malocclusion.
  Interventions: Device: Conventional facemask appliance
- Group 2 (Modified 3D printed facemask) (Experimental): Modified facemask appliances will be used for growing patients who have Cl. III malocclusion.
  Interventions: Device: Modified 3D printed facemask

INTERVENTIONS:
Device: Modified 3D printed facemask — modified 3D printed customized maxillary protraction facemask will be used for growing patients who have Cl. III malocclusion, hyrax expansion appliance and applying an elastic force of 300-500 gram per side for 12-14 hours per day. Treatment time 9 months.
  Arms: Group 2 (Modified 3D printed facemask)
Device: Conventional facemask appliance — Conventional facemask appliance will be used for growing patients who have Cl. III malocclusion, hyrax expansion appliance and applying an elastic force of 300-500 gram per side for 12-14 hours per day. Treatment time 9 months.
  Arms: Group 1 (Conventional facemask)

SUMMARY:
A randomized clinical trial to introduce a modified 3D printed customized maxillary protraction facemask and evaluate its efficacy in comparison with the conventional maxillary protraction facemask therapy in correction of Class III malocclusion of young patients

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two parallel arms. The patients will be randomly divided into two groups, group one: conventional facemask appliance will be used while group two, the modified facemask appliances. Lateral cephalometric x-ray, Study models, photographs, and patient questionnaire will be taken before starting the treatment (T0) and at the end of treatment (T1). The effectiveness of the two appliances will be assessed and measured comparing patient's records before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal and dental relationships: skeletal class III with retrognathic maxilla and normal mandible with overjet < 0 mm.
2. Concave profile with normal lower facial height (clinically and radiographically).
3. Good oral health free from caries and periodontal problems at the start of treatment.

Exclusion Criteria:

1. Previous history of orthopedic and/or orthodontic treatment.
2. Patients with vertical growth pattern or backward mandibular rotation tendency.
3. Patients with gross facial asymmetry.
4. Patients with cleft lip and palate and/or craniofacial syndrome
5. Patients with bad oral habit.
6. Active periodontal disease.
7. Previous history of TMJ signs or symptoms

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Dentoskeletal and soft tissue changes | (T0) before starting the treatment and (T1) after 9 months of treatments.
  Cephalometric analysis will be perfomed by measured different skeletal and soft tissue points in degrees at two time (T) intervals, (T0) before starting the treatment and (T1) at 9 months after treatment.

SECONDARY OUTCOMES:
Skeletal and soft tissue changes | (T0) before starting the treatment and (T1) after 9 months of treatments.
  Skeletal changes by comparing the changes of SNA, SNB and ANB angles in degrees using cephalometric x-rays at two time intervals, (T0) before starting the treatment and (T1) after 9 months of treatments.
Dental changes | (T0) before starting any treatment and (T1) after 9 months of treatments
  Dental changes will be evalauted by comparing over jet changes in millimeters assessed using study models.at two time intervals, (T0) before starting the treatment and (T1) after 9 months of treatments.

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - College of Dentistry-University of Baghdad, Baghdad, Al-Rusafa
  - Mushriq Abid, Baghdad

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdulkareem GB, Cobourne MT, Abid M. The effectiveness of novel 3D printed customized facemask appliance for treatment of class III malocclusion: a randomized clinical trial. Eur J Orthod. 2025 Oct 16;47(6):cjaf075. doi: 10.1093/ejo/cjaf075. PMID 41121454